CLINICAL TRIAL: NCT00086606
Title: A Phase II, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Oral Food Challenge Trial of Xolair (Omalizumab) in Peanut Allergy
Brief Title: A Safety and Efficacy Study of Xolair in Peanut Allergy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: Q2788g
Record Dates: First submitted 2004-07-06; First posted 2004-07-09 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Allergy
Keywords: Peanut
MeSH Terms: conditions — Hypersensitivity | interventions — Omalizumab

INTERVENTIONS:
Drug: Xolair (omalizumab)

SUMMARY:
This is a 38-week, randomized, double-blind, placebo-controlled, parallel group trial of approximately 150 patients who have a history of immediate hypersensitivity reaction to peanut protein.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of acute peanut allergy
* The patient meets the Xolair dosing table eligibility criteria by having a serum baseline IgE level between 30 and 1300IU/mL, and a body weight between 20 and 150 kilograms
* The patient is six to 75 years of age
* The patient reacts to peanut flour but not wheat (placebo) flour during the first Oral Food Challenge (OFC)
* The patient has a positive skin prick test to peanut or detectable serum peanut-specific IgE level
* The patient is able to swallow capsules

Exclusion Criteria:

* Have FEV1 value <80% predicted or any clinical features of moderate persistent asthma, as defined by the NHLBI guidelines
* Have other significant medical conditions (e.g., liver, gastrointestinal, kidney, cardiovascular, pulmonary disease, or blood disorders), which, in the opinion of the Investigator, make the subject unsuitable for induction of food reactions
* Have a history of allergy to wheat protein
* Have previously been exposed to monoclonal antibody treatment

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2004-06; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yamo Deniz, M.D., Study Director — Genentech, Inc.
Locations (1):
- Trial Information Support Line, Denver, Colorado, United States